CLINICAL TRIAL: NCT05905328
Title: Phase 1B/2A Study of CTO1681 for the Prevention and Treatment of Cytokine Release Syndrome in Patients With Diffuse Large B-Cell Lymphoma Receiving Chimeric Antigen Receptor T-Cell Therapy
Brief Title: Study of CTO1681 for the Prevention and Treatment of CRS in DLBCL Patients Receiving CAR T-Cell Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CytoAgents, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTA-2101
Record Dates: First submitted 2023-04-28; First posted 2023-06-15 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cytokine Release Syndrome
Keywords: Cytokine release syndrome; Cytokine storm; Hypercytokinemia; Immunotoxicity; CAR T-cell therapy
MeSH Terms: conditions — Cytokine Release Syndrome

STUDY DESIGN:
Intervention Model Description: The Phase 1b portion of the study is an open-label, dose-escalating, safety and pharmacokinetic (PK) study of multiple ascending doses of CTO1681 in patients with Diffuse Large B-cell Lymphoma who receive commercially available CD19-directed CAR T-cell therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CTO1681 30 μg Total Daily Dose (Experimental): Participants receive 10 μg CTO1681 orally 3 times daily (total daily dose of 30 μg) for 15 days.
  Interventions: Drug: CTO1681 10 μg
- CTO1681 60 μg Total Daily Dose (Experimental): Participants receive 20 μg CTO1681 orally 3 times daily (total daily dose of 60 μg) for 15 days.
  Interventions: Drug: CTO1681 20 μg
- CTO1681 90 μg Total Daily Dose (Experimental): Participants receive 30 μg CTO1681 orally 3 times daily (total daily dose of 90 μg) for 15 days.
  Interventions: Drug: CTO1681 30 μg

INTERVENTIONS:
Drug: CTO1681 10 μg — Administered 3 times daily for 15 days (initial cohort).
  Arms: CTO1681 30 μg Total Daily Dose
Drug: CTO1681 20 μg — Administered 3 times daily for 15 days (successive cohort).
  Arms: CTO1681 60 μg Total Daily Dose
Drug: CTO1681 30 μg — Administered 3 times daily for 15 days (successive cohort).
  Arms: CTO1681 90 μg Total Daily Dose

SUMMARY:
This is an interventional study to evaluate the use of CTO1681 in preventing or reducing CAR T-cell-induced toxicities like cytokine release syndrome (CRS). This study will enroll adult patients with DLBCL who are scheduled to receive CD19-directed CAR T-cell therapy.

The first phase of the study will be open label with dose escalation. Participants will start taking CTO1681 just prior to receiving their CAR T-cell therapy and continue to take the study drug three times daily for a total of 15 days.

DETAILED DESCRIPTION:
The first phase of the study will be an open-label, dose escalation, safety assessment in a group of patients, and will also collect data to investigate the potential benefit of CTO1681, initiated prior to CAR T-cell therapy, in preventing or reducing certain toxicities or side effects associated with CAR T-cell therapy, such as cytokine release syndrome (CRS).

Participants will start taking CTO1681 just prior to receiving their CAR T-cell therapy and continue to take the study drug three times daily for a total of 15 days.

Participants will provide blood samples at specified points throughout the study. In addition, urine samples, ECGs, scans, and other medical evaluations will be performed that are associated with the CAR T-cell therapy and/or necessary to verify study eligibility. Participants will be monitored for safety and efficacy for 43 days, and then will have follow-up to continue to monitor for safety and monitor for tumor response for up to 6 months for phase 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Undergone leukapheresis and is scheduled to receive protocol-specified commercially available CD19-directed CAR T-cell therapy (axicabtagene ciloleucel or lisocabtagene maraleucel) for DLBCL without corticosteroid prophylaxis for CRS and/or ICANS. Patients eligible for study must have relapsed or refractory DLBCL after at least one prior line of systemic therapy.
3. Met all inclusion criteria for CAR T-cell therapy per institutional guidelines.
4. Adequate organ function defined as:

   1. Estimated Creatinine Clearance per Cockroft Gault formula ≥ 60 mL/min.
   2. Serum alanine aminotransferase/aspartate aminotransferase ≤ 2.5 × ULN.
   3. Total bilirubin ≤ 1.5 × ULN.
   4. Left ventricular ejection fraction ≥ 40% on echocardiogram or multigated acquisition and no clinically significant pericardial effusion.
   5. Platelets ≥ 50,000/mm3.
   6. Absolute neutrophil count > 1000/μL.
   7. Absolute lymphocyte count > 100/μL.
5. Documented measurable lymphoma disease adequate to judge by Lugano Criteria.
6. Eastern Cooperative Oncology Group performance status 0 to 1.
7. Female participants of childbearing potential and all male participants must agree to use Investigator-approved methods of birth control while on study drug and for 30 days thereafter.
8. Patients who are willing to provide written informed consent before the predose procedures, or patients who have a legal representative capable of providing informed consent on their behalf.

Exclusion Criteria:

1. Any cytotoxic chemotherapy within 14 days prior to leukapheresis.
2. Clinically significant malabsorption syndromes and swallowing difficulties which are inadequately controlled with medication (eg, odynophagia, dysphagia, gastroesophageal reflux disease) as per Investigator assessment.
3. Grade 2 or greater electrolyte imbalance, per CTCAE v5.0:

   1. Potassium < 3.0 or > 5.5 mmol/L
   2. Sodium < 130 or > 150 mmol/L
   3. Calcium < 8.0 or > 11.5 mg/dL
   4. Magnesium < 0.5 or > 1.23 mmol/L
4. Clinically significant ECG abnormality at Screening or Baseline (Day -1), including but not limited to, a confirmed QTcF value > 470 msec. Patients to be excluded included those with QTcF readings that are borderline or difficult to interpret because of a condition such as bundle branch block, or in those where the end of the T wave is difficult to measure. This also includes any Grade 2 or greater conduction block disorder, atrial, or ventricular arrythmia.
5. History of clinically significant arrhythmia and/or requiring anticoagulation/antiplatelet treatment at therapeutic dose.
6. Any clinically significant (ie, active) cardiovascular disease, including cerebral vascular accident/stroke (< 6 months before enrollment), myocardial infarction (< 6 months before enrollment) or unstable angina, and congestive heart failure ≥ New York Heart Association Classification Class III.
7. Uncontrolled thromboembolic events or recent severe hemorrhage within the last 6 months.
8. Known history of any bleeding disorder.
9. Requirement for ongoing therapeutic doses of anticoagulant therapy, antiplatelet or fibrinolytic agents (low molecular weight heparin prophylaxis is allowed).
10. Baseline systolic blood pressure <100 mmHg.
11. History of autoimmune disease/ graft versus host disease requiring immunosuppressive therapy within the last 2 years. However, physiologic steroids (prednisone equivalent) may be given at a dose of 5 mg or less.
12. Patients who, in the opinion of the Investigator, would be unlikely to comply with study procedures or are otherwise unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 6 months following start of treatment
  AEs graded by CTCAE v5.0

SECONDARY OUTCOMES:
Incidence of CRS (any grade) | 6 months following the start of treatment
  CRS graded by ASTCT Consensus Grading
Incidence of ICANS (any grade) | 6 months following the start of treatment
  ICANS graded by ASTCT Consensus Grading
Incidence of hospitalizations | 6 months following the start of treatment
  Unplanned hospitalizations
Use of other anticytokine therapies | 6 months following the start of treatment
  Use of cytokine mitigating therapies other than CTO1681
Proinflammatory cytokine levels | 6 months following the start of treatment
  Concentration of proinflammatory cytokines in the blood
Concentration of CTO1681 | Baseline, Day 0, Day 2, Day 4, Day 6, Day 13
  Concentration of CTO1681 in the blood
CAR T-cell concentration in blood | 6 months following the start of treatment
  Concentration of CAR T-cell measured using ddPCR
CAR T-cell antitumor response | 6 months following the start of treatment
  Antitumor response assessment using the Lugano Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Bertolino, MD, PhD, MBA, Study Chair — CytoAgents, Inc.
Locations (6):
- United States (6):
  - University of California, Irvine - Chao Family Comprehensive Cancer Center, Orange, California
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Duke Cancer Institute, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No